CLINICAL TRIAL: NCT06962319
Title: A Multicentre Open-label, Non-inferiority Adaptive Platform Randomised Controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Antimalarials for the Treatment of Uncomplicated Malaria in the First Trimester of Pregnancy: Master Protocol
Brief Title: Safety of Antimalarials in the FIRst trimEster
Acronym: SAFIRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Malaria Research and Training Center, Mali International Center of Excellence in Research, University of Sciences, Techniques, and Technologies of Bamako, Mali (Unknown); KEMRI Centre for Global Health Research (CGHR), Kisumu, Kenya (Unknown); Clinical Research Unit of Nanoro (CRUN), Institut de Recherche en Sciences de la Santé (Unknown); Medicines for Malaria Venture (co-sponsor) (Unknown); US Centers for Disease Control and Prevention (CDC), Division of Parasitic Diseases & Malaria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-036; MMV_SAFIRE_24_01 (Other: Co-Sponsor identifier - Medicines for Malaria Venture)
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Malaria, Pregnancy; Malaria, Antepartum; Malaria (Uncomplicated)
Keywords: Malaria; Pregnancy; First trimester; antimalaria; artemether-lumefantrine; Adaptive Platform Trial
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: This is a Phase IIIb, multicentre, open-label, randomised, non-inferiority, Bayesian sequential adaptive platform clinical trial to investigate the efficacy, safety and tolerability of multipleantimalarial treatment arms simultaneously or sequentially in pregnant women in the first trimester of pregnancy with uncomplicated P. falciparum malaria.
  The study will be conducted in several phases, starting with an 'Initial' Phase consisting of a 3-arm trial, followed potentially by additional phases when new intervention arms are added. Any additional study arms added in the future will be described in the accompanying Intervention Specific Appendix (ISA[s]) and submitted for ethical and regulatory approvals. This open-ended trial continuously evaluates new antimalarials without a set end date, adapting to emerging treatments and research priorities in malaria during pregnancy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pyronaridine-artesunate (PA) (Experimental): PA is the latest registered ACT and is currently the only commonly used ACT singled out by WHO not to be used in the first trimester because of the lack of any safety data when the guidelines were reviewed. PA is currently seeing a rapid expansion of its use in Africa.
  Thus, PA is likely to be widely used in women of childbearing age in the coming years.
  Interventions: Drug: Pyronaridine-artesunate (PA)
- Dihydroartemisinin-piperaquine (DP) (Experimental): DP is an ACT widely used for the treatment of malaria and is registered in at least 30 malariaendemic countries, including Kenya, Mali and Burkina Faso. DP is also widely used in areas with multidrug-resistant P. falciparum and P. vivax in Southeast Asia. In Papua, Indonesia, DP was introduced as first-line treatment in 2006 in the general population, including in the 2nd and 3rd trimesters of pregnancy. DP is effective in reducing recurrent malaria and improving pregnancy outcomes in the second and third trimesters, offering significant benefits over quinine-based regimens. WHO includes DP as a recommended ACT for treating malaria in the second and third trimesters but emphasises the need for more safety data in the first trimester. The slower elimination of piperaquine that contributes to the longer duration of post-treatment prophylaxis relative to AL and the simplicity of the three-day treatment regimen (once daily as opposed to twice daily with AL).
  Interventions: Drug: dihydroartemisinin-piperaquine (DP)
- Artemether-lumefantrine (Active Comparator): Artemether-lumefantrine (AL) will serve as the first standard of care control arm in this platform trial comparing newer antimalarials. AL is the only drug recommended as first-line treatment for uncomplicated malaria in the first trimester of pregnancy, as per the World Health Organisation's 2022 updated guidelines. Other artemisinin-based combination therapies (ACTs) are only recommended if AL is unavailable.
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine (DP) — Weight-based dosing of 3 (<60kg), 4 (6-80kg) or 5 (>80 kg) 40/320 mg tablets of dihydroartemisinin-piperaquine given once daily for 3 days
  Arms: Dihydroartemisinin-piperaquine (DP)
Drug: Pyronaridine-artesunate (PA) — Weight-based dosing of 2 (24-<45 kg), 3 (45-<65kg), or 4 (>=65 kg) 180/60 mg tablets of pyronaridine-artesunate, once daily for 3 days.
  Arms: Pyronaridine-artesunate (PA)
Drug: Artemether-lumefantrine — 1 x 80/480 or 4 x 20/120 mg tablets of artemether-lumefantrine, given twice daily, approximately 8 hours apart for 3 days
  Arms: Artemether-lumefantrine

SUMMARY:
The SAFIRE study aims to find effective treatments with acceptable safety for malaria in early pregnancy, a particularly sensitive time for the adverse consequences of malaria in pregnancy for both mother and baby. Currently, WHO recommends the antimalarial drug artemether-lumefantrine (AL) for the treatment of uncomplicated malaria in the first trimester of pregnancy. Other promising treatments are being rolled out in malaria-endemic countries for use in adults and children and data on current exposures in the first trimester are limited and insufficient to support a recommendation. This is due to the fact that pregnant women are often excluded from clinical trials to protect fetuses, unintentionally depriving them of newer, potentially better treatments. Instead, they often received older, less effective drugs. The International Council for Harmonisation (ICH E21) and stringent regulatory authorities (e.g. EMA, FDA and MHRA) now encourage pregnant women to be included in well-designed studies to ensure they can safely benefit from medical advances.

This study will compare AL with the newer antimalarial drugs that have shown no significant safety concerns in laboratory studies, accidental use during early pregnancy, or trials in later pregnancy stages. The main goal is to see if these new drugs work as well as AL in treating malaria and are safe for the mother, her pregnancy and the developing baby. The newer antimalarials being tested also offer additional benefits to pregnant women, such as preventing new malaria infections for longer after treatment than the current standard treatment (AL). Also, they can be taken just once a day instead of twice daily, like AL. A simpler dosing schedule could improve adherence to the study medication, meaning women are more likely to take the full course of treatment as prescribed. This, in turn, enhances its effectiveness in real-world settings. Future antimalarials to be tested will include those with improved resistance profiles, offering more effective options for combating drug-resistant strains.

SAFIRE uses a special "Bayesian Adaptive Platform Trial" (APT) design. This open-ended approach allows researchers to add new interventions under the same protocol, leveraging the existing trial network with infrastructure. The use of a common protocol with innovative adaptive statistical design allows the trial to stop early if it becomes clear that the new drugs are unsafe.

This multi-centre trial will be conducted in several countries in Africa where malaria is very common. Women will be randomly assigned to receive either AL or one of the new treatments. Participants will be seen daily for 4 days, then weekly for 6 weeks to assess the response to treatment, and then monthly until delivery. Their health and outcomes will be closely monitored during and after pregnancy. Newborns will be followed for 6 months. An independent data safety and monitoring board (DSMB) will regularly monitor safety data as it accumulates. By finding more treatment options, this study could improve care for pregnant women with malaria and lead to better health for mothers and babies in areas where malaria is widespread. The results will help inform global health policies and potentially change how we treat malaria in early pregnancy.

DETAILED DESCRIPTION:
Background: Malaria in pregnancy remains a substantial public health concern in endemic regions, with first-trimester infections being particularly harmful. The World Health Organization (WHO) now recommends artemether-lumefantrine (AL), an artemisinin-based combination therapy (ACT), as the first-line treatment for uncomplicated malaria in the first trimester of pregnancy, replacing quinine. This recommendation followed a comprehensive review of observational data on inadvertent first-trimester exposures from pregnancy exposure registries, which showed that initial concerns about the teratogenicity of artemisinin derivatives raised by preclinical studies and animal models did not apply to human pregnancies.

Several other highly effective ACTs are used in sub-Saharan Africa, a trend likely to increase rapidly as part of WHO's multiple first-line strategies. Moreover, novel treatments that show promise against resistant strains and may potentially impede their emergence or spread could become available. SAFIRE aims to efficiently generate evidence on the safety and efficacy of antimalarials for treating uncomplicated malaria in the first trimester. Each of the antimalarials to be evaluated in this SAFIRE trial should meet the following criteria:

* Registered antimalarial product for the treatment of uncomplicated malaria or at minimum, confirmation of a favourable benefit/risk ratio for the treatment of uncomplicated malaria in a confirmatory Phase III program in children or adults with P. falciparum infection
* No teratogenic concerns in preclinical studies

In the case of antimalarials with a teratogenic signal in preclinical studies:

* No significant safety concerns in women inadvertently treated with these drugs in the first trimester (from observational studies and/or pregnancy exposure registries),

Ideally, no significant safety, tolerability and efficacy concerns in clinical trials during the second and third trimesters of pregnancy would be preferred.

Justification: It took over two decades to accumulate sufficient evidence for WHO to recommend AL for use in the first trimester. There is an urgent need to expedite this process and provide informed guidance to health care providers and mothers on other potentially effective and safe antimalarials, especially in the context of the increased threat of resistance against AL. Furthermore, stringent regulatory authorities now encourage more research involving pregnant women.

Objectives: The primary efficacy objective in the initial phase of this adaptive platform trial is to confirm the efficacy of alternative antimalarials in pregnant women in the first trimester with uncomplicated malaria by demonstrating non-inferiority to the current standard of care with AL. The key safety objective is to assess their non-inferiority compared with AL in terms of safety regarding pregnancy outcomes.

Study design: SAFIRE is a multicentre, open-label, randomised, non-inferiority, adaptive platform trial (APT). The rationale for a non-inferiority approach is that if these newer drugs prove to be non-inferior to AL in terms of efficacy and safety, they offer secondary advantages such as longer post-treatment prophylaxis or simpler dosing regimens (once instead of twice daily for 3 days). These benefits could improve treatment adherence and effectiveness in real-world settings.

The study employs a Bayesian adaptive design, allowing for interim analyses and potential early stopping for safety. The rule for making decisions during interim analysis is to stop enrolment to a new intervention arm if there is more than an 85% chance that the hazard ratio for the safety endpoint exceeds 1.1 (the non-inferiority margin) relative to the standard of care. These frequent interim analyses for safety will allow for the early stopping of the trial arm if safety concerns arise and enable more efficient use of resources and timely decision-making based on accumulating evidence.

The adaptive platform trial design evaluates multiple interventions and uses a shared control group, reducing administrative burden and allowing efficient participant allocation. It provides a flexible framework for introducing new treatment arms, which is ideal for assessing multiple promising antimalarials for first-trimester use.

SAFIRE is an open-ended trial that continuously evaluates new antimalarials without a set end date, adapting to emerging treatments and research priorities in malaria during pregnancy.

The protocol uses a modular design with a master protocol outlining the overall framework and intervention-specific appendices (ISAs) for each antimalarial. This approach enables efficient addition or removal of treatment arms without full master protocol revision, enhancing flexibility and responsiveness.

Methods: Pregnant women in their first trimester (≤13 weeks' gestation) with confirmed uncomplicated Plasmodium falciparum malaria will be randomly assigned to receive either the standard of care with artemether-lumefantrine (AL) or a newer antimalarial. The details of the newer antimalarials, corresponding sample sizes, and allocation ratio are described in ISAs. The primary efficacy endpoint is PCR-adjusted adequate clinical and parasitological response (ACPR) by day 42. The key safety endpoint is a composite of fetal loss or major congenital anomalies. Secondary efficacy endpoints include PCR-unadjusted cure rates (i.e, the cumulative rate of women without recurrent malaria infection due to treatment failure or reinfection), serving as a proxy for the duration of post-treatment prophylaxis.

Collaboration and funding: The initial phase of the study is co-sponsored by the Liverpool School of Tropical Medicine (LSTM) and the Medicines for Malaria Venture (MMV) and is funded by Global Health EDCTP3, the EU, UKRI, and SERI of the Swiss Confederation. As this is an open-ended platform trial, additional sponsors and funders may be added in the future as new treatment arms are incorporated.

Ethical considerations and governance: The trial adheres to stringent ethical standards, including obtaining informed consent from all participants and providing close monitoring for adverse events. An independent Data Safety Monitoring Board will monitor the safety data as they accumulate with predefined stopping rules.

Significance: SAFIRE is designed to inform WHO policy. By expanding the range of safe and effective treatment options, SAFIRE has the potential to improve the management of malaria in early pregnancy, an important period for the developing placenta and fetus, and contribute to better maternal and child health outcomes in endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 weeks and <14 weeks (13-6/7 weeks inclusive) gestation from the last menstrual period (LMP) as assessed by echography
* Microscopy confirmed P. falciparum mono or mixed infections, regardless of symptoms.
* Emancipated minor and aged ≥16 years
* Haemoglobin ≥ 7 g/dL
* Residence within the health facility catchment area
* Willingness to adhere to study requirements and to deliver the baby at the local health facility
* Willingness to adhere to study requirements and to deliver the baby at the local health facility

Exclusion Criteria:

* Known allergy to any of the study drugs
* History of known pregnancy complications or poor obstetric history, such as repeated miscarriages, stillbirths, or eclampsia
* History or presence of major illnesses likely to influence pregnancy outcome
* Known HIV positive
* Any significant illness at the time of screening requiring hospitalisation, including severe malaria
* Intent to move out of the study catchment area before delivery or planned delivery out of the catchment area
* Recent (2 weeks) treatment with antimalarials or antimicrobials with antimalarial activity (chloroquine, AL, DP, PA, SPAQ, ASAQ, MQAS, azithromycin, clindamycin, tetracycline, quinolones, cotrimoxazole and SP)
* Twin/multiple pregnancy detected
* Non-viable pregnancy confirmed by ultrasound or doppler
* Known history or evidence of clinically significant cardiovascular disorders or family history of sudden death or congenital long QT syndrome or current co administration of other drugs that might contribute to a prolonged QTc interval or cause "Torsades de Point"
* Chronic medical condition requiring frequent medications (e.g., TB, suspected hepatic lesions, liver disease, sickle cell disease, diabetes, epilepsy, asthma and hypertension)
* Prior randomisation in this study during the current pregnancy

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1510 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
ACPR | Day 42
  PCR-adjusted adequate clinical and parasitological response (ACPR) by Day 42

SECONDARY OUTCOMES:
Efficacy - ACPR Day 28 | Day 28
  PCR-adjusted Adequate clinical and parasitological response by Day 28

OTHER OUTCOMES:
Primary safety endpoint - delivery | Delivery
  A composite endpoint of miscarriage, stillbirth, or major congenital anomalies

CONTACTS AND LOCATIONS:
Overall Officials: Fieko ter Kuile, MD, Principal Investigator — Liverpool School of Tropical Medicine; Kassoum Kayentao, MD, Principal Investigator — Universite des Sciences, des Techniques et des Technologies de Bamako; Stephanie Dellicour, PhD, Principal Investigator — Liverpool School of Tropical Medicine; Hellen Barsosio, MD, Principal Investigator — KEMRI Centre for Global Health Research (CGHR); Innocent Valea, PhD, Principal Investigator — Institut de Recherche en Sciences de la Santé (IRSS); Myriam El Gaaloul, PharmD, Principal Investigator — Medicines for Malaria Venture
Locations (3):
- Clinical Research Unit of Nanoro (CRUN), Institut de Recherche en Sciences de la Santé, Direction Régionale de l'Ouest (IRSS-DRO), Nanoro, Burkina Faso
- KEMRI Centre for Global Health Research (CGHR), Kisumu, Kenya
- Malaria Research and Training Center, University of Sciences, Techniques, and Technologies of Bamako (USTTB),, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified dataset of the complete patient-level data
Time Frame: No later than one year after the publication of the trial results - no end date decided
Access Criteria: Through a data sharing repository platform such as WWARN.

REFERENCES:
- See also: Project website — https://safire-consortium.org/